CLINICAL TRIAL: NCT06195540
Title: RIVACAST : RIVAroxaban Versus Low-molecular Weight Heparinin Patients With Lower Limb Trauma Requiring Brace or CASTing
Brief Title: RIVAroxaban Versus Low-molecular Weight Heparin in Patients With Lower Limb Trauma Requiring Brace or CASTing
Acronym: RIVACAST
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 49RC21_0376; 2023-509905-62-00 (EU CTIS Number)
Record Dates: First submitted 2023-12-22; First posted 2024-01-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Venous Thromboembolism; Deep Vein Thrombosis; Pulmonary Embolism; Lower Limb Trauma; Thromboprophylaxis; Immobilisation
Keywords: Emergency department; direct oral anticoagulant; rivaroxaban; Low-Molecular-weight heparin; randomized control trial; Prevent VTE
MeSH Terms: conditions — Venous Thromboembolism; Venous Thrombosis; Pulmonary Embolism; Emergencies | interventions — Rivaroxaban; Dalteparin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Open label with blind assessment of study's outcomes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rivaroxaban arm (Experimental)
  Interventions: Drug: Rivaroxaban 10 MG
- Low-molecular-weight heparin arm (Active Comparator): Treatment with LMWH is the standard-of-care in this population of lower limb trauma patients at risk of thrombosis.
  The control group is therefore the group of patients who receive prophylactic anticoagulant treatment with LMWH for the duration of immobilization (i.e. until full mobilization with weight-bearing).
  Interventions: Drug: Low Heparin Molecular Weight

INTERVENTIONS:
Drug: Rivaroxaban 10 MG — Administration of rivaroxaban 10 mg once daily to prevent venous thromboembolic events in patients with trauma to a lower limb.
  Consecutive patients with lower limb trauma and a TRiP(cast) score ≥ 7 are assessed for possible participation in the study. At the inclusion visit, if the patient meets the study's selection criteria, the investigator provides oral and written information (information letter written in a language the patient can understand) and answers any questions the patient may have. Depending on randomisation, the patient will receive either LMWH or rivaroxaban. The dose is rivaroxaban 10 mg orally once a day (no dosage adjustment).
  Treatment is started in the emergency department and continued at home for the duration of the immobilisation (i.e. until mobilisation with weight-bearing). The duration of treatment will be determined by the physician.
  Arms: Rivaroxaban arm
Drug: Low Heparin Molecular Weight — Administration of standard prophylactic anticoagulant treatment with LMWH for the duration of immobilisation (i.e. until full mobilisation with weight-bearing). Consecutive patients with lower limb trauma and a TRiP(cast) score ≥ 7 are assessed for possible participation in the study. At the inclusion visit, if the patient meets the study's selection criteria, the investigator provides oral and written information (information letter written in a language the patient can understand) and answers any questions the patient may have. Depending on randomisation, the patient will receive either LMWH or rivaroxaban. The dose of LMWH is free, given according to local practices and national recommendations.
  Treatment is started in the emergency department and continued at home for the duration of the immobilisation (i.e. until mobilisation with weight-bearing). The duration of treatment will be determined by the physician.
  Arms: Low-molecular-weight heparin arm

SUMMARY:
Lower limb trauma requiring immobilization is a very frequent condition that is associated with an increased risk of developing venous thromboembolism (VTE). The TRiP(cast) score has been developed to provide individual VTE risk stratification and help in thromboprophylactic anticoagulation decision. The recent CASTING study had confirmed that patients with a TRiP(cast) score <7 have a very low risk of VTE and could be safely manage without prophylactic treatment. Conversely, patients with a score ≥ 7 have a high-risk of VTE and require a prophylactic anticoagulant treatment. Low molecular weight heparins (LMWH) have been shown to be effective in this indication. However, in the CASTING study, the 3-month symptomatic VTE rate was 2.6% in this subgroup despite LMWH prophylactic treatment. This result suggests that LMWH are not sufficiently effective in this particular subgroup of high-risk patients. Direct oral anticoagulants, and in particular rivaroxaban, may be an effective and safe alternative to LMWH. In the PRONOMOS study, comparing LMWH with rivaroxaban in patients who had undergone non-major lower limb surgery, the relative risk of symptomatic VTE was 0.25 (95% CI = 0.09 - 0.75) in favor of rivaroxaban 10mg. No significant increase in bleeding was found. In addition, as LMWH treatment requires subcutaneous daily injections, the use of rivaroxaban may positively impact patients' quality of life as well as being effective in medico-economic terms.

The aims of this study are to demonstrate that rivaroxaban is at least as effective, easier to use and more efficient than LMWH in patients with trauma to the lower limb requiring immobilisation and deemed to be at risk of venous thromboembolism (TRiP(cast) score ≥ 7). High-risk patients are randomized to receive either rivaroxaban or LMWH. They are followed up at 45 days and 90 days to assess the occurrence of thrombotic events or bleeding, as well as their satisfaction with the treatment received.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 or over ;
* Consultation in an emergency department of a participating centre;
* Trauma to the lower limb requiring rigid or semi-rigid orthopaedic immobilisation;
* Expected duration of orthopaedic immobilisation of at least 2 weeks;
* TRiP(cast) score ≥ 7 ;
* Patient affiliated to or benefiting from a social security scheme;
* Patient with prior informed consent.

Exclusion Criteria:

* Patient that have to be hospitalized after emergency department for other reason than lower limb trauma
* Active bleeding or high risk of bleeding,
* Known contraindication to rivaroxaban or LMWH;
* Taking any anticoagulant or antiplatelet agent before the trauma (only antithrombotic authorised: aspirin < 325mg/d);
* Pregnant or breastfeeding woman;
* Any factor making 3-month follow-up impossible; 6. Patient subject to a legal protection measure, Imprisonment 7. Participation in any interventional study which modifies patient care or could influence study evaluation criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1424 (Estimated)
Dates: Start 2024-07-19 (Actual); Primary Completion 2026-11-19 (Estimated); Study Completion 2026-11-19 (Estimated)

PRIMARY OUTCOMES:
Rate of symptomatic venous thromboembolic events (45 days non-inferiority) | 45 days
  The primary endpoint is the rate of symptomatic venous thromboembolic events (including deep vein thrombosis and/or pulmonary embolism and/or PE-related death) within 45 days (+/- 5 days) of inclusion.
  Symptomatic VTE is defined as follows:
  * Deep venous thrombosis (DVT) of the lower limbs: DVT confirmed by a non-compressible venous segment on compression ultrasound or by a filling defect on CT venography. Symptomatic proximal and distal DVTs will be taken into account.
  * Symptomatic pulmonary embolism documented by thoracic angioscan, high probability planar lung scan, SPECT scan, pulmonary angiography or by the combination of documented proximal deep vein thrombosis and thoracic symptomatology suggestive of pulmonary embolism.
  * PE-related deaths according to the ISTH (International Society of Thrombosis and Haemostasis) definition All events will need to be confirmed by the randomisation group's blinded clinical events adjudication committee.

SECONDARY OUTCOMES:
Patient self reported treatment satisfaction | 45 days
  The outcome is patient self-reported treatment satisfaction using the Anti-Clot Treatment Scales (ACTS) assessed at 45 days (+/- 5 days).
Rate of symptomatic venous thromboembolic events (90 days superiority) | 90 days
  This secondary outcome is the cumulative rate of symptomatic venous thromboembolism (i.e., deep venous thrombosis and/or pulmonary embolism) within the 90 days (± 7 days) after the inclusion.
  The definition of symptomatic VTE is the same as the primary outcome.
Cumulative rates of major bleeding and of non-major clinically relevant bleeding (90 days) | 90 days
  The cumulative rates of major bleeding and of non-major clinically relevant bleeding at 90 days (± 7 days).
  Major bleeding is defined according to the International Society of Thrombosis and Haemostasis (ISTH) criteria and includes:
  * Any bleeding resulting in death
  * Symptomatic bleeding in a critical organ including intracranial, intraspinal, intraocular, retroperitoneal, intra-articular, pericardial bleeding and muscle bleeding resulting in compartment syndrome,
  * Symptomatic bleeding resulting in a decrease in the haemoglobin concentration of at least 2g/dL or resulting in the transfusion of at least two packs of blood red cells.
  Clinically Relevant Non-Major Bleeding is defined as:
  - Any bleeding requiring hospitalisation or a medical intervention including temporary withholding of anticoagulant treatment to stop the bleeding.
Incremental cost-utility ratio (rivaroxaban efficiency 45 days) | 45 days
  The incremental cost-utility ratio (costs per quality-adjusted life year (QALY) gained) assessed at 45 days after inclusion. Health-related quality of life will be collected using EQ-5D-5L self-administered questionnaires at each scheduled follow-up at 45 days (±/- 5). Resources consumed will be taken from french national Health Data System.
Incremental cost-utility ratio (rivaroxaban efficiency 90 days) | 90 days
  The incremental cost-utility ratio (costs per quality-adjusted life year [QALY] gained) assessed at 90 days after inclusion. Health-related quality of life will be collected using EQ-5D-5L self-administered questionnaires at each scheduled follow-up at at 90 days (± 7). Resources consumed will be taken from french national Health Data System.

CONTACTS AND LOCATIONS:
Overall Officials: Delphine Douillet, Doctor, Study Director — Angers University Hospital
Locations (35):
- France (35):
  - Agen-Nerac Hospital, Emergency Department, Agen
  - Angers University Hospital, Emergency department, Angers
  - Argenteuil hospital, Emergency department, Argenteuil
  - Arpajon Hospital, Emergency Department, Arpajon
  - Caen University hospital, Emergency department, Caen
  - Tours University Hospital, Emergency department, Chambray-lès-Tours
  - Cholet Hospital, Emergency department, Cholet
  - Clermont-Ferrand University Hospital, Emergency department, Clermont-Ferrand
  - Simone Veil Hospital, Emergency Department, Eaubonne
  - Eure-Seine Hospital, Emergency Departement, Évreux
  - Grenoble University Hospital, Emergency Department, Grenoble
  - La Rochelle Hospital, Adult emergency departement, La Rochelle
  - Le Mans Hospital, Emergency department, Le Mans
  - Limoges University hospital, Emergency department, Limoges
  - Edouard Herriot University Hospital, Emergency Department, Lyon
  - Marseille University Hospital, Emergency department, Marseille
  - Melun Hospital, Emergency Department, Melun
  - Montpellier University Hospital, emergency department, Montpellier
  - Nantes University Hospital, Emergency department, Nantes
  - Nice University Hospital, Emergency department, Nice
  - Niort Hospital, Emergency Department, Niort
  - Lariboisière hospital, emergency department, Paris
  - Saint-Antoine Hospital, Emergency department, Paris
  - La Pitié-Salpétrière Hospital, Emergency Department, Paris
  - Cochin Hospital, Emergency department, Paris
  - St-Joseph Hospital, Emergency Department, Paris
  - HEGP, Emergency Department, Paris
  - Bichat Hospital, Adult Emergency department, Paris
  - South Lyon University Hospital, Emergency department, Pierre-Bénite
  - Poitiers University Hospital, Emergency department, Poitiers
  - Rennes University Hospital, Emergency department, Rennes
  - Rouen University Hospital, Emergency Department, Rouen
  - Strasbourg University Hospital, Emergency Department, Strasbourg
  - Toulouse University Hospital, Emergency Department, Toulouse
  - Vannes Hospital, Emergency Department, Vannes

IPD SHARING:
Plan to Share IPD: Undecided